CLINICAL TRIAL: NCT02710188
Title: A Phase 1 Relative Bioavailability Study in Healthy CYP2D6 Intermediate (IM) and Extensive Metaboliser (EM) Subjects, Designed to Evaluate the Pharmacokinetic (PK) Profile of HTL0009936 Following Single Dose Administration of Modified Release (MR) Prototype Formulations
Brief Title: Relative Bioavailability Study in Healthy Subjects to Evaluate the Pharmacokinetics of HTL0009936 After One Dose of Prototype Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9936-104; 2015-004921-16 (EudraCT Number)
Record Dates: First submitted 2016-03-02; First posted 2016-03-16 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HTL0009936 modified release (MR) Formulation (Experimental): Intervention: 5 different modified release formulations of HTL0009936, as a single dose
  Interventions: Drug: HTL0009936 modified release
- HTL00009936 immediate release (IR) fasted (Active Comparator): Intervention: 1 immediate release formulation of HTL0009936, as a single dose in the fasted state
  Interventions: Drug: HTL0009936 immediate release

INTERVENTIONS:
Drug: HTL0009936 modified release — HTL0009936 modified release
  Arms: HTL0009936 modified release (MR) Formulation
Drug: HTL0009936 immediate release — HTL0009936 immediate release
  Arms: HTL00009936 immediate release (IR) fasted

SUMMARY:
The purpose of this study is to find a modified release oral tablet formulation for this drug, which will be safe and well tolerated.

DETAILED DESCRIPTION:
The aim of the study is to develop a modified release oral tablet formulation that maintains plasma concentrations within the target therapeutic range, and is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males & females
* Aged 18 to 65 years
* Body mass index of 18.0 to 35.0 kg/m2
* CYP2D6 (intermediate or extensive metabolizer)

Exclusion Criteria:

* Subjects with a resting heart rate (HR) >90 bpm, and/or systolic blood pressure (BP) >150 mmHg, and/or diastolic BP >90 mmHg
* Subjects with QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms (males) or >470 ms (females)
* Personal or family history of long QT syndrome or sudden death
* Subjects who are CYP2D6 (poor or ultra-rapid metabolizer)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Tlag | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of the elapsed time from dosing at which HTL0009936 was first quantifiable in a concentration vs time profile (Tlag).
Frel | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of relative bioavailability (Frel) of HTL0009936 MR prototype formulations compared to the IR reference formulation and, if applicable, MR prototype formulations in the fed state compared to fasted state.
Tmax | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of the elapsed time from dosing at which the maximum observed HTL0009936 concentration (Cmax) was apparent (Tmax)
Cmax | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of Cmax.
Concentration of HTL0009936 at 6 hours post dose (C6) | 6 hours post dose
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of HTL0009936 concentration at 6 hours post-dose (C6)
AUC (0-last) | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of the area under the concentration versus time curve from time zero to the last measurable concentration (AUC(0-last))
AUC (0-inf) | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of the area under the concentration versus time curve from time zero to extrapolated to infinity (AUC(0-inf)).
AUC%extrap | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of percentage of AUC(0-inf) extrapolated beyond last measured time point (AUC%extrap).
Lambda-z | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of the slope of the apparent elimination phase (Lambda-z).
T1/2 | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of the apparent elimination half-life (T1/2).
Dose normalized AUC | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. In addition, if different dose levels of the same prototype are administered, dose normalized AUC (AUC/D) will be calculated.
Dose normalized Cmax | 14 weeks
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. In addition, if different dose levels of the same prototype are administered, dose normalized Cmax (Cmax/D) will be calculated.
Concentration of HTL0009936 at 12 hours post dose (C12) | 12 hours post dose
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of HTL0009936 concentration at 12 hours post-dose (C12)
Concentration of HTL0009936 at 24 hours post dose (C24) | 24 hours post dose
  The PK profiles of HTL0009936 Modified release oral prototype formulations in healthy CYP2D6 IM and EM subjects. Calculation of HTL0009936 concentration at 24 hours post-dose (C24)

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MBChB, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No